CLINICAL TRIAL: NCT02857725
Title: Sun Protection Factor (SPF) Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18300
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreen Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPF evaluation (Experimental): Subjects with good health as determined from the CRO Subject History Form (SHF) and Fitzpatrick Skin Type I, II and/or III were considered for SPF testing.
  Interventions: Drug: BAY 987517; Drug: SPF 15 Control

INTERVENTIONS:
Drug: BAY 987517 — Single dose application of two (2) mg/cm² of test product. Each 50 cm² test site area requires 100 mg of a product to obtain a standard 2 mg/cm² test application.
Drug: SPF 15 Control — Single dose application of two (2) mg/cm² of test product. Each 50 cm² test site area requires 100 mg of a product to obtain a standard 2 mg/cm² test application.

SUMMARY:
Evaluation of the effectiveness of a sunscreen product by determining its Sun Protection Factor (SPF) on the skin of human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of an age of 18 to 70 years inclusive;
* Fitzpatrick Skin Type I, II and/or III for SPF testing;
* Good health as determined from the CRO Subject History Form (SHF);
* Signed and dated Informed Consent Form;
* Signed and dated Health Insurance Portability and Accountability Act (HIPAA) Form;
* An unambiguous minimal erythema dose (MED).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2015-06-09 (Actual); Study Completion 2015-06-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of water resistant SPF in accordance to 21 CFR (Code of Federal Regulations) 207.327 | 16-24 h post exposure

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Union, New Jersey, United States